CLINICAL TRIAL: NCT00277186
Title: A Randomized Controlled Prospective Study to Examine the Effectiveness of a New Evidence Based Arthroplasty Care Model for Patients With Severe Degenerative Joint Disease (DJD) of the Hip or Knee in Alberta
Brief Title: Alberta Hip and Knee Replacement Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Bone and Joint Health Institute (Other)
Collaborators: Alberta Medical Association (Other); Calgary Health Region (Other); David Thompson Health Region (Unknown); Capital Health Region (Unknown); Alberta Health & Wellness (Other Government)
Responsible Party: Alberta Bone and Joint Health Institute, Alberta Bone and Joint Health Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARTH-00001
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
Keywords: Arthroplasty; Health services research; Intent to treat; Randomized; Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Patients entering new care continuum
  Interventions: Other: New Care Continuum
- Control (Active Comparator): Patient enter existing conventional approach
  Interventions: Other: New Care Continuum

INTERVENTIONS:
Other: New Care Continuum — Patient experience surgery through newly designed arthroplasty continuum

SUMMARY:
The study aims to determine if a New Arthroplasty Care Model, established on evidence-based medicine and best practices, will improve patient outcomes and improve cost effectiveness for patients with severe degenerative joint disease of the hip or knee in Alberta

DETAILED DESCRIPTION:
The Alberta Orthopaedic Society through its Arthroplasty Service Design Working Group has, after carefully reviewing the existing conventional approach to arthroplasty care, developed what they believe could be a much improved new evidence based arthroplasty care model. This model represents how ideally a patient would access and receive health services across the complete continuum of care. In addition, wherever possible, evidence gathered from the literature and from "known best practices" has been utilized to develop standards related to access, wait times, clinical quality, resource use and health outcome measures. Where no evidence or "known best practices" exist, a standard that best support achieving other known standards are being developed. This new evidence based arthroplasty model seeks to significantly minimize and where possible, eliminate all the current gaps and barriers to arthroplasty care.

This study will seek to prove that the new evidence based arthroplasty model will deliver improved patient outcomes with improved cost effectiveness. Once proven, it is anticipated that this new evidence based arthroplasty model will become the standard of care in Alberta, and a model for other jurisdictions to use in their health service re-designs

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient is able to provide written consent

Exclusion Criteria:

* Patient has previously undergone arthroplasty of the same hip or knee (revision)
* Patient has a surgical date scheduled for arthroplasty
* Patient requires a hip resurfacing procedure or an oxford knee
* Patient has a concurrent medical condition that would contraindicate the patients' ability to participate fully in the study procedures, including terminal conditions such as chronic obstructive pulmonary disease, end stage renal disease, heart failure, malignancy with an anticipated life expectancy of ≤ 2 years
* Patient has senile dementia or Alzheimer's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3434 (Actual)
Dates: Start 2005-04; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
health related quality of life scores | 3 month and 12 months post-surgery

SECONDARY OUTCOMES:
health resource utilization | 3 month and 12 months post-surgery
wait time | Pre-surgery
safety | 3 month and 12 months post-surgery
cost utility | 3 month and 12 months post-surgery
patient satisfaction | 3 month and 12 months post-surgery
provider satisfaction | 3 month and 12 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Frank, MD, Principal Investigator — University of Calgary; Bill Johnston, MD, Principal Investigator — University of Alberta
Locations (1):
- Alberta Bone and Joint Health Institute, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Gooch K, Marshall DA, Faris PD, Khong H, Wasylak T, Pearce T, Johnston DW, Arnett G, Hibbert J, Beaupre LA, Zernicke RF, Frank C. Comparative effectiveness of alternative clinical pathways for primary hip and knee joint replacement patients: a pragmatic randomized, controlled trial. Osteoarthritis Cartilage. 2012 Oct;20(10):1086-94. doi: 10.1016/j.joca.2012.06.017. Epub 2012 Jul 11. PMID 22796513